CLINICAL TRIAL: NCT01200173
Title: Effect of the Consumption of a Fermented Milk on Common Infections in Children Aged 3-6 Years, Attending Day Care Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NU206
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Common Infectious Diseases
Keywords: Probiotic - Lactobacillus casei DN-114 001 - dairy; product - infections - children

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 = Tested product (Active Comparator)
  Interventions: Other: 1-Fermented dairy product containing the probiotic Lactobacillus casei DN-114 001 (Actimel®)
- 2 = Control product (Sham Comparator)
  Interventions: Other: 2-Non fermented dairy product (control)

INTERVENTIONS:
Other: 1-Fermented dairy product containing the probiotic Lactobacillus casei DN-114 001 (Actimel®)
  Arms: 1 = Tested product
Other: 2-Non fermented dairy product (control)
  Arms: 2 = Control product

SUMMARY:
This multicentric, randomized, double-blind and controlled study aims to examine the effect of a fermented dairy product containing the probiotic Lactobacillus casei DN-114 001 (Actimel® = tested product) on the incidence of respiratory and gastro-intestinal common infectious diseases (cumulated number of infections during the intervention period: primary criteria) in children aged 3-6 years, attending day care centers.Volunteers received either 200g/day of tested product (N=300) or control product (N=299) for 3-months, followed by a 1-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subject whose parents/legal guardians had given written informed consent,
* Male or female, aged 3 to 6 years (upper bound excluded),
* Attending day-care centres or preschools 5 days a week in the Moscow area,
* Subject found medically healthy (in particular, free of respiratory and GI tract symptoms),
* Subject who appreciated dairy products and multi-fruit flavour.

Exclusion Criteria:

* Subject whose parents were not reading and writing Russian, or not understanding informed consent or study protocol.
* Subject with allergy or hypersensitivity to milk proteins or dairy foods components (ex: lactose, milk proteins), or with any known food or respiratory allergy.
* Subject presenting a severe evolutive or chronic pathology (Ex: cancer, tuberculosis, Crohn disease, cirrhosis, multiple sclerosis, Type I diabetes…) or any past or actual health condition that could interfere with the outcome of the study (Ex: HIV, Chemotherapy, malabsorption, ulcer, celiac disease, failure to thrive…).
* Subject having experienced any infectious disease during the last 7 days.
* Subject with current diarrhoea or constipation Subject who was frequently using laxatives or who had been using laxatives during the week prior his participation to the study.
* Subject who was under artificial nutrition, had gastro-intestinal surgery or any intervention requiring general anaesthesia the last 2 months prior to his participation to the study.
* Subject with special medicated diet (obesity, anorexia, metabolic pathology, nutritional complementation…) or with eating disorders (anorexia, bulimia…).
* Subject currently receiving, or who had received during the last months, systemic treatment or topical treatment likely to interfere with evaluation of the study parameters: antibiotics, antiseptics, antifungal, corticoids, vaccines, anti-histaminic molecules, non-corticoid antiinflammatory substances, immunosuppressant treatment…
* Subject already enrolled in another clinical study, or currently under an exemption period from a previous study.
* Subject in a situation which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Institution "Federal research center of pediatric hematology, oncology and imunology", Moscow, Russia

REFERENCES:
- [Derived] Prodeus A, Niborski V, Schrezenmeir J, Gorelov A, Shcherbina A, Rumyantsev A. Fermented Milk Consumption and Common Infections in Children Attending Day-Care Centers: A Randomized Trial. J Pediatr Gastroenterol Nutr. 2016 Nov;63(5):534-543. doi: 10.1097/MPG.0000000000001248. PMID 27168455